CLINICAL TRIAL: NCT01626586
Title: Adjustment and Self-Management Intervention Groups for Youth With Type 1 Diabetes Mellitus
Brief Title: Diabetes Adolescent and Family Group Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Marquette University (Other)
Responsible Party: Principal Investigator, Jessica Kichler, Ph.D., C.D.E., Principal Investigator, Children's Hospital Medical Center, Cincinnati
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-1200
Record Dates: First submitted 2012-06-19; First posted 2012-06-25 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Youth; Family; Group Therapy; Type 1 Diabetes Mellitus; Self-Management
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Psychotherapy, Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group Therapy (Experimental): This study includes having an initial assessment completed; participating in a 6 session group therapy intervention over a 7 week time period; and returning at 2 and 4 months after group therapy intervention for "booster" follow-up sessions. During the group intervention sessions, the parent group and the youth group will each meet for about 45 minutes and then the families will come together to work on family goals for the last 15 to 20 minutes.
  Interventions: Behavioral: Group Therapy
- Individual Arm (Active Comparator): This study includes having an initial assessment completed; participating in a 6 session individual therapy intervention over a 7 week time period; and returning at 2 months after the individual therapy intervention for the "booster" follow-up session. During the individual intervention sessions, the youth and the parents will each meet for about 45 minutes and then the families will come together to work on family goals for the last 15 to 20 minutes.
  Interventions: Behavioral: Group Therapy
- Recently Diagnosed Arm (Active Comparator): This study includes enrolling patients with Type 1 Diabetes, who are recently diagnosed (<1 year) to participate in a 4 session group therapy intervention over a 4 week time period; and returning at 2 months after the last group session for the "booster" follow-up session. During the group sessions, the youth and the parents will each meet for about 45 minutes and then the families will come together to work on family goals for the last 15-20 minutes.
  Interventions: Behavioral: Group Therapy

INTERVENTIONS:
Behavioral: Group Therapy — Self-management Diabetes Protocol: Successful adjustment to daily diabetes management requires a wealth of clinical knowledge, solid problem-solving and coping skills to deal with the physical, social and emotional factors associated with caring for and living with a chronic illness, and motivation to take care of one's health.

SUMMARY:
In this research study the investigators want more about how being in a group about diabetes helps your family versus individual treatment. The investigators are now asking youth with recently diagnosed (<1 year) diabetes and their parents to be in the research, because the investigators want to see if this diabetes group and/or individual therapy is helpful to your coping, adjustment, and family communication about diabetes.

DETAILED DESCRIPTION:
The purpose of this research study is to find out what effects the Group Therapy Project has on parents and child's management of Type 1 Diabetes Mellitus (T1DM) from both a group versus an individual therapy modality. We want to start a group and individual therapy program that looks at youth and family adjustment and coping at the Cincinnati Children's Hospital with patients who have T1DM. There has been research before on this group therapy and we want to look at it in a "typical" clinical setting at Cincinnati Children's Hospital for both group and individual therapy, including recently diagnosed patients (<1 year). This research is being done to understand how a peer and family-based group versus individual therapy can be helpful by looking at survey data as well as medical data before and after participating in the diabetes therapy program. This information will help us further develop prevention and intervention programs for other youth with T1DM and their families.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 1 Diabetes,
* Aged 10.0 - 17.9 years of age,
* At least one parent/caregiver to participate with them,
* Diagnosed for at least 6 months for the Group and the Individual Arms.
* Diagnosed for <1 year for the Recently Diagnosed Arm

Exclusion Criteria:

* Potential participants will be excluded if:

  * They have a co-existing diagnosis of mental retardation, pervasive developmental disorder, substance abuse, eating disorders, psychosis, or other acute psychiatric or medical needs, such as suicidality
  * They are not fluent in the English language.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Diabetes-related Outcomes | 8 years
  Diabetes-related improvements for the youths and their parents (e.g., diabetes responsibility, adherence, and parent-child interactions) from baseline to post-treatment, maintenance of these changes over the 2 and 4 month follow-up.

SECONDARY OUTCOMES:
Diabetes-related medical outcome data | 8 years
  Medical improvements for youth (e.g., HbA1c) pre- to post-treatment and maintained at 6 months after the last booster session. Decreased health care utilization for the youth (e.g., emergency room visits and inpatient hospitalizations) pre- to post-treatment and maintained at 6 months after the last booster session.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Kichler, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States